CLINICAL TRIAL: NCT04314336
Title: The Economic Impact of Clinical Pharmacist Involvement in the Public Procurement for Medicines and in the Work of the Drug and Therapeutics Committee, Single-centre, Cost-minimisation Study
Brief Title: The Economic Impact of Clinical Pharmacist Involvement in the Public Procurement for Medicines and in the Drug and Therapeutics Committee
Status: Completed | Type: Observational
Sponsor: Bjelovar General Hospital (Other)
Responsible Party: Principal Investigator, Eugen Javor, MPharm, Clinical Pharmacist, Bjelovar General Hospital
Other Study IDs: 1520192020
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Rationalization
Keywords: Rationalization; Clinical Pharmacist; Public Procurement for Medicines; Drug and Therapeutics Committee
MeSH Terms: interventions — Pharmaceutical Preparations; Pharmacy and Therapeutics Committee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Public procurement — Cost minimisation study through public procurement
Drug: Drug and Therapeutics Committee — Cost minimisation analysis of results of the drug and therapeutics committee before and after clinical pharmacist involvement

SUMMARY:
The investigators have performed cost-minimisation analysis and compared the expenses based on the plan for public procurement (without clinical pharmacist involvement) for drugs with the results of public procurement based on the revised plan for public procurement by the clinical pharmacist. The plan for public procurements was based on the 1 year quantity for each medicine used by the hospital in the previous year, based on the latest deliverable prices at the time of extracting the data to workbook for MS Excel program (ver. 2002, Microsoft, Redmond, WA, USA).

The investigators have performed cost-minimisation analysis and compared the expenses for all received requests for medicines to the drug and therapeutics committee (DTC) for a decision in the 1 year period, before and after involvement of clinical pharmacist in the committee work. The expenses were based on approval decisions in the 1 year period for approval time period. The denial decisions were also calculated and reported. The denial period calculated in rationalisation of expenses were based on 1 year treatment period.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the hospital (inhospital patients)

Exclusion Criteria:

* None

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inhospital patients, all patients receiving any medicine during their stay in the hospital within 1 year period.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Reducing prices of medicines | 1 year
  Reduce prices of medicines in percentage, since different countries and hospitals have various budgets and medicine prices

SECONDARY OUTCOMES:
Rationalization of expenses | 1 year
  Rationalization of expenses through rquests for medicines sent to Drug and Therapeutics Committee

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital Bjelovar, Bjelovar, Croatia

IPD SHARING:
Plan to Share IPD: No